CLINICAL TRIAL: NCT02995980
Title: Pilot Study of Dual-energy (DE) Contrast-enhanced (CE) Digital Mammography to Detect Breast Cancer in Patients With Increased Breast Density (Breast Imaging-Reporting And Data System (BI-RADS) Category c or d)
Brief Title: Study of Dual-energy (DE) Contrast-enhanced (CE) Digital Mammography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Rachael Lancaster, MD, MD, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: F141210004
Record Dates: First submitted 2016-03-20; First posted 2016-12-19 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer
Keywords: breast cancer screening; dense breasts; dual-energy contrast-enhanced digital mammography
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Contrast enhanced mammography vs standard digital mammogram (Experimental): Contrast-enhanced spectral mammography for the detection breast cancer .
  Interventions: Device: Dual-Energy Contrast-Enhanced (DECE) mammography; Device: digital mammography

INTERVENTIONS:
Device: Dual-Energy Contrast-Enhanced (DECE) mammography — Contrast mammography
  Other Names: Contrast-enhanced spectral mammography (CESM); Contrast-enhanced mammography
Device: digital mammography — routine digital mammography
  Other Names: full field digital mammography

SUMMARY:
This is a feasibility study to evaluate dual-energy (DE) contrast-enhanced (CE) digital mammography to detect breast cancer in patients with increased breast density (BI-RADS category c or d). Eligible patients will be invited to have full-field digital mammography and dual-energy (DE) contrast-enhanced (CE) digital mammography to compare accuracy of the imaging methods for the detection of breast cancer.

DETAILED DESCRIPTION:
This is a feasibility study to evaluate dual-energy (DE) contrast-enhanced (CE) digital mammography to detect breast cancer in patients with increased breast density (Breast Imaging-Reporting And Data System category c or d). Eligible patients will be invited to have full-field digital mammography and dual-energy (DE) contrast-enhanced (CE) digital mammography to compare accuracy of the imaging methods for the detection of breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. At least 19 years old
3. Glomerular filtration rate> 60
4. Heterogeneously or extremely dense breasts (BI-RADS category c or d).

Exclusion Criteria:

1. History of iodinated contrast allergy
2. Pregnant or lactating as determined by routine standard practice
3. Personal history of breast cancer
4. History of prior breast excisional biopsy (Patients with a history of core needle biopsy will not be excluded)
5. History of prior breast reduction mammoplasty surgery
6. History of prior breast augmentation surgery
7. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2015-11; Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi R Umphrey, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The Kirklin Clinic, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Contrast Enhanced Mammography vs Standard Digital Mammograpm: Contrast-enhanced spectral mammography for the detection breast cancer .
  Dual-Energy Contrast-Enhanced (DECE) mammography: Contrast mammography
Period: Overall Study
Arm/Group | Contrast Enhanced Mammography vs Standard Digital Mammograpm
Started | 128
Completed | 114
Not Completed | 14
Not completed — Lost to Follow-up | 14

BASELINE CHARACTERISTICS:
Population: 114 patients completed both mammograms
Groups:
- Contrast Enhanced Mammography vs Standard Digital Mammograpm: Contrast-enhanced spectral mammography for the detection breast cancer .
  DECE mammography: Contrast mammography
Arm/Group | Contrast Enhanced Mammography vs Standard Digital Mammograpm
Number analyzed (Participants) | 128
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 100
  >=65 years | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 100
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Accuracy of Contrast Mammography
Description: •The primary endpoint of this study is to determine the accuracy of DE CE mammography when compared to full field digital mammography (FFDM) in patients with increased breast density (Breast Imaging-Reporting And Data System (BI-RADS) category c or d breast density).
Time Frame: 1 year
Population: Consented 128 patients, 114 patients completed both mammograms
Measure: Number (95% Confidence Interval); unit: percentage of accuracy
Groups:
- Contrast Enhanced Mammography: Contrast-enhanced spectral mammography for the detection breast cancer .
  DECE mammography: Contrast mammography
- Standard Digital Mammogram: Full field digital mammography for the detection breast cancer
  digital mammography: routine digital mammography
Arm/Group | Contrast Enhanced Mammography | Standard Digital Mammogram
Number analyzed (Participants) | 114 | 114
percentage of accuracy | 100 [29 to 100] | 67 [9 to 99]

2. Primary Outcome: Number of Participants With Cancer Detected
Description: •The primary endpoint of this study is to detect the presence of cancer using DE CE mammography when compared to full field digital mammography (FFDM) in patients with increased breast density (BI-RADS category c or d breast density).
Time Frame: 1 year
Population: Consented 128 patients, 114 patients completed both mammograms
Measure: Count of Participants; unit: Participants
Arm/Group | Contrast Enhanced Mammography | Standard Digital Mammogram
Number analyzed (Participants) | 114 | 114
Participants | 3 | 2

3. Secondary Outcome: Number of Call Backs With Contrast Mammography
Description: •The patients identified for additional imaging based on unconfirmed findings.
Time Frame: 1 year
Population: Consented 128 patients, 114 patients completed both mammograms
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Contrast Enhanced Mammography | Standard Digital Mammogram
Number analyzed (Participants) | 114 | 114
percentage of participants | 10 [5 to 17] | 11 [6 to 19]

ADVERSE EVENTS:
Time Frame: Adverse events will be recorded on the CRFs up to 30 days after administration of the last dose of study treatment.
Arm/Group | Contrast Enhanced Mammography vs Standard Digital Mammograpm
All-Cause Mortality (participants affected / at risk) | 0/128
Serious Adverse Events (participants affected / at risk) | 0/128
Other Adverse Events (participants affected / at risk) | 0/128

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/80/NCT02995980/Prot_SAP_ICF_000.pdf